CLINICAL TRIAL: NCT00254696
Title: Association of Antibiotic Utilization Measures and Control of Extended-spectrum-lactamases (ESBLs)
Brief Title: Study Evaluating Antibiotic Utilization Measures and Control of Extended-Spectrum-Lactamases (ESBLs)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0910X-101462
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Bacterial Infection
Keywords: bacterial infection
MeSH Terms: conditions — Bacterial Infections

INTERVENTIONS:
Drug: Extended-Spectrum-Lactamases (ESBLs)

SUMMARY:
* To determine the value of using piperacillin/tazobactam in reducing the cases of ESBL producing E. coli or K. pneumoniae colonization and infection.
* To determine the acquisition rate of ESBL producing E. coli or K. pneumoniae, both pre and post intervention in the selected medical centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted or transferred to the ICU/pulmonary/hematology units.
* Patients of either sex, 18 years of age or older

Exclusion Criteria:

* Pregnant and nursing women. Female of childbearing potential without using any birth control methods. Female of childbearing potential using oral contraceptives during study period. (Note: penicillin and beta-lactamase inhibitors may prevent oral contraceptives from working properly, increasing the chance of pregnancy).
* Patients who have the contraindications of using Tazocin (pipercillin/tazobactam)

Other exclusions apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Actual)
Dates: Start 2004-06; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Acquisition rate of ESBL producing E. coli or K. pneumoniae at the end of phase I (pre-intervention) and phase II (last 3 months)

SECONDARY OUTCOMES:
Infection rate of ESBL producing E. coli or K. Pneumoniae at the end of phase I (pre-intervention) and phase II (last 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For China medinfo@wyeth.com